CLINICAL TRIAL: NCT02580968
Title: Study of Key Electro-acupuncture Technique on Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 643857003534
Record Dates: First submitted 2015-07-30; First posted 2015-10-20 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Migraine
Keywords: Electroacupuncture therapy; Migraine; Acupuncture Therapy
MeSH Terms: conditions — Migraine Disorders | interventions — Flunarizine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- electro-acupuncture (Experimental): 100hz, 2min. electro-acupoint: LI4(Large Intestine4) with LV3(Liver3).5times a week. lasting for 4 weeks.
  Interventions: Device: electro-acupuncture
- routin medicine (Active Comparator): one tablet of flunarizine hydrochloride tablet per day. lasting for 20days
  Interventions: Drug: flunarizine hydrochloride

INTERVENTIONS:
Device: electro-acupuncture — electro-acupuncture on acupoints according to the traditional syndrome diagnosis.once per day, for 20 days.
  Arms: electro-acupuncture
Drug: flunarizine hydrochloride — flunarizine hydrochloride ，10mg/day，for 20 days。
  Other Names: flunarizine
  Arms: routin medicine

SUMMARY:
A random controlled trail to evaluate the efficacy of migraine standard electroacupuncture formula, and to analysis the regulation of the intensity-effects and to observe the peripheral NO, CGRP and NF-кB expression level of migraine patients after electroacupuncture treatment.

DETAILED DESCRIPTION:
acupuncture group(group A): treated by acupuncture for 20 days, 1 time per day control group(group B): treated by FlunarizineHydrochloride for 20 days, 1 table per day.

ELIGIBILITY:
Inclusion Criteria:

* met the diagnostic criteria for migraine; suffering from migraine attacks; migraine attacks for more than 5 days per month, and lasts for 3 months; voluntarily join this study with informed consents.

Exclusion Criteria:

* other systemic, neurological and psychiatric disorders; headache caused by other diseases; not treatment compliance during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-03; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Migraine Disability Assessment Questionnaire (MIDAS) | 20 days
  a scientifically reliable and valid measure of migraine disability that can improve communication between patients and physicians, assess migraine severity and act as an outcome measure to monitor treatment efficacy

SECONDARY OUTCOMES:
The medical outcomes study 36-item short-form health survey(SF-36) | 20 days
  A 36-item short-form (SF-36) was constructed to survey health status in the Medical Outcomes Study
peripheral Nitrogen Monoxide(NO) protein expression | 20 days
  marker
peripheral Calcitonin gene related peptide(CGRP) protein expression | 20 days
  marker
peripheral Nuclear factor-kappa B(NF-кB) protein expression | 20 days
  marker
Visual Analogue Scale (VAS) to assess pain | 20 days
  Visual Analogue Scale (VAS) were applied to measure pain in patients

CONTACTS AND LOCATIONS:
Overall Officials: Jian Pei, Ph.D, Study Director — Longhua Hospital
Locations (1):
- Longhua Hospital,Shanghai University of Traditional Chinese Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No